CLINICAL TRIAL: NCT03203616
Title: Multicenter, Non-randomised, Open-label, Single Agent Phase II Study to Determine the Clinical Benefit of Trastuzumab Emtansine (T-DM1) in HER2-positive Metastatic Breast Cancer Patients With Brain Metastasis
Brief Title: Kadcyla In pAtients With bRAin Metastasis
Acronym: KIARA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: As most HER2+ patient develop brain mets while on/after having received TDM1, it has proven to be an insurmountable challenge to recruit patients
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IJB-BC-TDM1BM-2016
Record Dates: First submitted 2017-04-24; First posted 2017-06-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Metastatic HER2-positive Breast Cancer With Brain Metastasis
MeSH Terms: interventions — Ado-Trastuzumab Emtansine; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kadcyla (T-DM1) (Experimental): trastuzumab emtansine given every 3 weeks at the standard dose (3.6 mg/kg) via intravenous infusion, until disease progression, intolerable toxicity or consent withdrawal. A median of 9 cycles per patient is expected
  Interventions: Drug: KADCYLA 160 MG Injection

INTERVENTIONS:
Drug: KADCYLA 160 MG Injection — Kadcyla 160Mg Powder for Injection: 3.6 mg/kg iv every 3 weeks
  Other Names: T-DM1; trastuzumab emtansine

SUMMARY:
Women with breast cancer often develop metastases in the brain. Currently, treatment of these metastases is difficult and relies on radiotherapy or surgery which often fail. Therefore, development of new methods of treatment for breast cancer with brain metastasis is very important. T-DM1 is a drug that is already in everyday use for a specific type of breast cancer called HER2-positive breast cancer. The objective of this study is to investigate whether T-DM1 is also effective in brain metastasis and can help patients to live longer and better

DETAILED DESCRIPTION:
This is a multicentre, non-randomised, open label, single arm, phase II study of T-DM1 in patients with metastatic breast cancer and with brain metastasis who have already failed at least one line of anti-HER2 therapy for systemic disease. The study sample is composed of 2 distinct cohorts of patients.

Cohort number 1 is composed of patients with asymptomatic or oligosymptomatic brain metastasis (single or multiple), measurable according to RECIST 1.1, who have not received any local therapy (neither surgery, radiosurgery nor whole brain radiotherapy) for brain metastasis.

Cohort number 2 is composed of patients with brain metastasis (single or multiple), measurable according to RECIST 1.1, previously treated with local therapy (surgery, radiosurgery or whole brain radiotherapy) and with radiologically confirmed brain progression, with a minimum period of 3 months between the end of local therapy and brain progression.

A total number of 110 are planned for screening, in order to enrol 97 patients. A minimum of 87 evaluable patients is necessary. Inclusion of patients in both cohorts will follow a two-stage Simon optimal design. During the study, both brain assessments via magnetic-resonance imaging (MRI) and systemic assessments with computerised tomography (CT) will be performed every 3 cycles (9 weeks) of therapy.

Study treatment consists of T-DM1, 3.6 mg/kg every 3 weeks. Patients will receive study medication until unacceptable toxicity, voluntary withdrawal from study treatment, disease progression, death or pregnancy, whichever occurs first. Patients who experience only progression in the brain and who receive local therapy may remain in the study until systemic progression (or any of the other reasons stated previously), at the investigator's discretion.

After the end of study treatment, all patients will have a safety visit within 30 days (+/- 7 days) from the last T-DM1 administration date. After the safety visit, according the reason of end of study treatment, the follow-up period will begin, as described below:

* If study treatment stopped due to progression of disease Patients will enter directly in survival follow-up. No visits are mandatory per protocol after the safety visit. Chart review and/or phone call to check if the patient is still alive are to be performed, every 6 months, in order to acquire data for the overall survival endpoint. Patients in survival follow-up who are of childbearing potential must be tested for pregnancy at 3 months and at 7 months after end of study treatment. These tests can be ordered by the investigator during regular out of study follow-up visits.
* If study treatment stopped for any other reason than progression (either toxicity or voluntary withdrawal from study treatment) Patients will enter first in efficacy follow-up after the safety visit and then in survival follow-up when progression disease is observed.

During efficacy follow-up, 9 weekly efficacy assessments continue according to the same timetable they would have followed had treatment interruption not occurred. This consists of imaging assessments (MRI and CT) and medical visits, as well as QoL evaluations. During this period, treatment is at the discretion of the local physician/investigator.

This follow-up is to continue until disease progression or until voluntary withdrawal of the patient from the study. In case this follow-up is impossible (due to patient refusing to perform assessments or other reasons), survival data can be collected every 6 months via chart review or telephone. Patients in follow-up who are of childbearing potential must be tested for pregnancy at 3 months and at 7 months after end of study treatment. Once a patient has progressed while on efficacy follow-up, they will enter into survival follow-up as per description above.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all these criteria in order to be eligible for the study:

General Criteria:

* Female patients (≥ 18 years);
* Histologically confirmed HER2-positive breast cancer patients (IHC 3+ and/or ISH positive);
* Patients should have previously received trastuzumab and a taxane, separately or in combination. Patients should have either received prior therapy for locally advanced or metastatic disease, or developed disease recurrence during or within six months of completing adjuvant therapy;
* At least one measurable brain metastasis as defined by RECIST 1.1 (≥ 10 mm);
* Any hormone receptor status;
* Predicted life expectancy > 3 months;
* Any previous anti-HER2 therapies are allowed, other than T-DM1;
* ECOG performance score 0-2;
* No significant cardiac history and a current LVEF ≥ 50%. LVEF should be determined within 21 days before enrolment;
* Adequate organ function, evidenced by the following laboratory results. Exams are to be performed at a maximum of 7 days before enrolment.

  * Absolute neutrophil count > 1,500 cells/mm3 without growth factor support (14 days after last peg-filgrastrim, 7 days for regular filgrastrim).
  * Platelet count > 100,000 cells/mm3 without transfusion 2 weeks prior assessment
  * Hemoglobin > 9 g/dL without transfusion 2 weeks prior assessment.
  * Aspartate aminotransferase and alanine aminotransferase < 2.5 x upper limit of normal (ULN).
  * Total bilirubin ≤ 1.5 x ULN unless the patient has documented Gilbert's syndrome, in which case direct (conjugated) bilirubin level needs to be within normal limits.
  * Serum alkaline phosphatase ≤ 2.5 x ULN. Patients with bone metastases: alkaline phosphatase ≤ 5 x ULN.
  * Serum creatinine < 2.0 mg/dL or < 177 μmol/L.
  * International normalized ratio (INR) and activated partial thromboplastin time or partial thromboplastin time < 1.5 ULN unless patient receiving anticoagulant therapy
* For women of childbearing potential a serum pregnancy test will be done up to 7 days before enrolment (and it must be negative) and an agreement to use one highly-effective form of non-hormonal contraception (true abstinence, vasectomy, oophorectomy/hysterectomy, IUD) or two effective forms of non-hormonal contraception (e.g., condoms plus spermicidal agent) at study entry (to be put in place within 2 weeks prior to enrolment), during the administration of T-DM1 and for 7 months after the last administration of T-DM1 will be obtained
* Signed informed consent obtained before any study-specific procedure;
* Able and willing to comply with the protocol; including the willingness to provide samples (primary if available and blood) for translational research.

Cohort 1 additional specific criteria:

* No corticosteroids at enrolment
* Oligosymptomatic or asymptomatic brain metastases not requiring immediate local therapy.

Cohort 2 additional specific criteria:

* Radiologically confirmed brain progression after previous local therapy (neurosurgery, radiosurgery to the brain, stereotactic radiotherapy to the brain, or whole brain radiotherapy) with at least 3 months between end of local therapy and brain progression.
* Decreasing corticosteroid dose or stable dose for at least one week prior to enrolment

Exclusion Criteria:

Patients who exhibit any of the following conditions at screening will be ineligible for admission into the study:

General Criteria:

* Single brain metastasis with indication of surgical resection
* Pregnant or breast-feeding women
* Documented leptomeningeal disease
* Having received any investigational therapy within ≤ 28 days or 5 half-lives at ICF signature, whichever is longer
* Having received hormonal therapy within 14 days of enrolment
* Having received trastuzumab within 21 days of enrolment
* Prior enrolment in a T-DM1-containing study, regardless of whether the patient received T-DM1 or not
* History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins or any component of the product.
* Current peripheral neuropathy of Grade ≥ 3 according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v.4.0.3
* History of other malignancy within the last 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other cancers with a similar outcome as those mentioned above.
* Current unstable ventricular arrhythmia requiring treatment.
* History of symptomatic congestive heart failure (CHF) (New York Heart Association [NYHA] Classes II-IV).
* History of myocardial infarction or unstable angina within 6 months prior to first study drug administration.
* Current dyspnoea at rest due to complications of advanced malignancy or currently requiring continuous oxygen therapy.
* Current severe, uncontrolled systemic disease other than cancer (e.g., clinically significant pulmonary, hypertension or metabolic disease)
* Concurrent, serious, uncontrolled infections or current known infection with HIV, active hepatitis B and/or hepatitis C.
* Major surgical procedure or significant traumatic injury within 28 days before enrolment or anticipation of the need for major surgery during the course of study treatment.
* Known contraindications for undergoing MRI or CT, including to receive contrast media,

Cohort 1 : additional specific criteria:

• Previous neurosurgery or radiotherapy (radiosurgery, stereotactic radiotherapy, whole brain radiotherapy) to the brain Cohort 2 : no additional specific criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Clinical Benefit (CB) | 9 weeks
  defined as complete response plus partial response plus stable disease in the brain, measured by RECIST 1.1, as determined by the local investigators.

SECONDARY OUTCOMES:
CB in the brain RECIST 1.1 | 9 weeks
  measured by RECIST 1.1 criteria, as determined by central evaluation
CB in the brain RANO | 9 weeks
  measured by RANO brain metastases criteria, as determined by the local investigators
General and cardiac-specific safety | up to 30 days after last treatment administration
  AEs and SAEs according NCI-CTCAE v4.03
CB: Systemic | 9 weeks
  defined as complete response plus partial response plus stable disease in non brain areas
CB: bi-compartmental | 9 weeks
  defined as complete response plus partial response plus stable disease in the whole body
Overall Response (OR) in the brain | 9 weeks
  defined as complete response plus partial response in brain
Overall Response (OR) systemic | 9 weeks
  defined as complete response plus partial response in non brain
Overall Response (OR) bi-compartmental | 9 weeks
  defined as complete response plus partial response in the whole body
Best Response (BR) in the brain | 1 year
  defined as the best obtained response in the brain
Best Response (BR) systemic | 1 year
  defined as the best obtained response in the non brain
Best Response (BR) bi-compartmental | 1 year
  defined as the best obtained response in the whole body
Brain Progression free survival (PFS) | 1 year
  defined as time between enrolment in the study and progression in the brain
Systemic PFS | 1 year
  defined as time between enrolment in the study and progression in areas other than the brain
Bi-compartmental PFS | 1 year
  defined as time between enrolment in the study and progression of disease
Duration of response in the brain | 1 year
  defined as time from documentation of tumour response in the brain (PR or CR) to disease progression in the brain
Duration of response systemic | 1 year
  systemic defined as time from documentation of non-brain tumour response (PR or CR) to non-brain progression
Duration of response bi-compartmental | 1 year
  Bi-compartmental defined as time between response and progression
Duration of Clinical Benefit (DCB) in the brain | 1 year
  defined as the time elapsed between determination of SD, PR or CR and determination of disease progression in the brain
Duration of Clinical Benefit (DCB) systemic | 1 year
  defined as the time elapsed between determination of SD, PR or CR and determination of systemic disease progression
Duration of Clinical Benefit (DCB) bi-compartmental | 1 year
  defined as the time elapsed between determination of SD, PR or CR and determination of bi-compartmental disease progression
Overall survival | 1 year
  defined as time between enrolment in the study and death
Quality of life | 1 year
  Quality of life will be assessed using the EORTC validated questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Evandro de Azambuja, MD, Study Chair — Jules Bordet Institute

IPD SHARING:
Plan to Share IPD: No